CLINICAL TRIAL: NCT04392180
Title: COA-APTIC Caregiver Concept Elicitation Study: A Qualitative Concept Elicitation Study to Identify Important Aspects of Pain Assessment, Treatment, and Response to Treatment in Children Who Are 0 to <3 Years of Age
Brief Title: COA-APTIC Caregiver Concept Elicitation Study
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pro00105117
Record Dates: First submitted 2020-05-14; First posted 2020-05-18 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2021-08

CONDITIONS: Pain Measurement
Keywords: acute pain; pediatrics
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregivers: Caregivers who care for a child that is both under 3 years of age and has experienced acute pain.
  This cohort will participate in a qualitative interview about pain assessment, treatment, and response to treatment in their child.
  Interventions: Other: Qualitative Interview

INTERVENTIONS:
Other: Qualitative Interview — There is no intervention as part of this study. Caregivers will participate in a qualitative interview over the phone or by video.

SUMMARY:
This is a concept elicitation study to identify important aspects of pain assessment, treatment, and response to treatment in children under than 3 years of age from a caregiver's perspective.

DETAILED DESCRIPTION:
The purpose of this study is to identify important endpoints and outcomes for use in pediatric trials for acute pain therapeutics in infants and young children from a caregiver's perception. Study team members will conduct phone-based qualitative interviews, using a semi-structured interview guide, with 42 primary caregivers of pediatric patients under 3 years of age who are experiencing or have experienced acute pain. Once participants give verbal consent, they will fill out a demographics form. Interviews will last about one hour and will address the participant's experience recognizing and managing their child's acute pain. The investigators will use these concept elicitation interviews to identify important aspects of acute pain assessment, treatment, and response to treatment in children who are under 3 years old. Interviews will be audio recorded and transcribed with participant permission. Transcripts or interviewer notes will be reviewed by two analysts and will be double coded until inter-rater reliability is reached by agreement of at least 80%. The study team will conduct a thematic analysis of the coded transcripts. This is a minimal risk study. All information will be kept confidential and information will be stored on a secure network which is only accessible to the study team.

ELIGIBILITY:
Inclusion Criteria:

1. Cares for a child who is both:

   * Between 0 and <3 years of age
   * Experiencing or has experienced acute pain in one of the following categories:
   * Malignant or non-malignant visceral or hematologic disease
   * Surgery (or other procedure)
   * Trauma or injury
   * Congenital conditions
2. Is over the age of 18 years old.
3. Can speak and understand English.
4. Is capable of and willing to provide informed consent for interview participation and to collect medical data from the child's medical record.

Exclusion Criteria:

1. Lack of access to a telephone or computer for interview
2. Has a child with acute pain that is extremely premature (less than 32 weeks gestation at the time of enrollment) and no other eligible child.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be caregivers of children 0 to <3 years old who have experienced acute pain. Eligible caregivers will be identified by Pediatric Trials Network sites across the United States. Eligible participants will be identified through recruitment for a pre-existing Pediatric Trials Network study called Pharmacokinetics and Safety of Anesthetics and Analgesics in Children and Adolescents.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Caregiver perspective on how to identify or recognize pain in children 0 to <3 years old. | 1 hour
  A 1-hour qualitative interview will be conducted and transcript or interviewer notes will be coded to assess how caregivers identify and recognize acute pain in infants and young children.
Caregiver perspective on how and when to intervene for acute pain in children 0 to <3 years old. | 1 hour
  A 1-hour qualitative interview will be conducted and transcript or interviewer notes will be coded to assess caregiver's perspective on how and when to treat acute pain in infants and young children.
Caregiver perspective on how to evaluate response to treatment for acute pain in children 0 to <3 years old. | 1 hour
  A 1-hour qualitative interview will be conducted and transcript or interviewer notes will be coded to assess how caregivers evaluate response to treatment for acute pain in infants and young children.
Caregiver perspective on important side effects of acute pain therapeutics in children 0 to <3 years old. | 1 hour
  A 1-hour qualitative interview will be conducted and transcript or interviewer notes will be coded to assess caregiver's perspective on important side effects of acute pain in infants and young children.

CONTACTS AND LOCATIONS:
Overall Officials: Bryce Reeve, PhD, Principal Investigator — Duke University; Kanecia Zimmerman, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside of the study team.